CLINICAL TRIAL: NCT06099080
Title: Open-Label Study of the Safety and Efficacy of SM-020 Gel 1.0% in Subjects With Dermatosis Papulosa Nigra
Brief Title: A Trial to Study the Safety and Efficacy of SM-020 Gel 1.0% in Subjects With Dermatosis Papulosa Nigra (DPN)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-216
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dermatosis Papulosa Nigra
MeSH Terms: conditions — Dermatosis Papulosa Nigra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SM-020 gel 1.0% (Experimental): Subjects will apply the investigational product twice daily for 4 consecutive weeks. Subjects will be followed for 12 weeks post final application for a total of approximately 16 weeks of required participation in the study.
  Interventions: Drug: SM-020 gel 1.0%

INTERVENTIONS:
Drug: SM-020 gel 1.0% — Subjects will apply the investigational product twice daily for 4 consecutive weeks. Subjects will be followed for 12 weeks post final application for a total of approximately 16 weeks of required participation in the study.

SUMMARY:
An open-label trial to explore the safety and efficacy of SM-020 gel 1.0% in subjects with Dermatosis Papulosa Nigra (DPN). Approximately 10 subjects will be enrolled with DPNs to apply SM-020 gel 1.0%. Each subject must have a minimum of 5 eligible DPNTLs with a diameter ≥2mm but ≤5mm. A maximum of 10 DPNs per subject will be targeted for treatment. Subjects will apply the investigational product twice daily for 4 consecutive weeks. Subjects will be followed for 12 weeks post final application for a total of approximately 16 weeks of required participation in the study. A total of 5-10 eligible Dermatosis Papulosa Nigra Target Lesions (DPNTLs) will be treated per subject.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to comprehend and willing to sign an informed consent form (ICF)
2. Must complete a signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of the subject's individually identifiable health information
3. Must be a male or female >18 years of age at the time of signing the informed consent form
4. Subject has Fitzpatrick Skin Type of 4, 5, or 6
5. Subject has a clinical diagnosis of Dermatosis Papulosa Nigra (DPN)
6. DPNTLs must:

   1. Have a minimum of 5 eligible facial DPNTLs. A maximum 10 DPNTLs will be targeted for treatment. An eligible DPNTL must have one or more clinical features throughout the entirety of the lesion: clustered, small (<5mm), waxy, warty, stuck-on, sharply demarcated, tan to black papules, milia-like cysts, on the cheeks and temples in people of color, particularly of African or Asian descent (Duffill, 2008).
   2. For subjects randomized for eligibility assessment with dermoscopy, DPNTLs must also have one or more of the following dermoscopy features throughout the entirety of the lesion: milia-like cysts, comedo-like openings, fissures/ridges, cerebriform surface (fat fingers)
   3. Have a diameter that is ≥2mm but ≤5mm
   4. Have a Physician's DPN Lesion Assessment Score (DPNLA) of > 2
   5. Be a discrete, well-defined, separate lesion
   6. Not be covered with hair which, in the Investigator's opinion, would interfere with the study gel treatment or the study evaluations
   7. Not be on the eyelids
   8. Not be within 5mm of the orbital rim
   9. Not be pedunculated
   10. Not be inflamed, irritated, or excoriated
7. Must be free of any known disease state or physical condition which, in the Investigator's opinion, might impair evaluation of any DPNTL or which exposes the subject to an unacceptable risk by study participation.
8. Must be willing and able to follow all study instructions and to attend all study visits.
9. Must be willing to have all partial or incompletely responding DPNTLs removed surgically by shave excision during the final visit.

Exclusion Criteria:

Exclusion Criteria Subjects meeting any of the following criterion will be ineligible and excluded from this study:

1. Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control (such as oral contraceptive pills (OCPs), Intrauterine devices (IUDs), birth control implants, vaginal rings, or injections) for the duration of the study.
2. DPN lesions that are clinically atypical and/or rapidly growing in size or number.
3. Presence of multiple eruptive DPN or SK lesions (sign of Leser-Trelat)
4. Current systemic malignancy.
5. Any use of the following systemic therapies within the specified period, or unwilling to meet the following washouts, prior to the Baseline visit and while on study:

   1. Retinoids; 180 days
   2. Chemotherapy; 180 days
   3. Immunosuppressive therapy; 28 days
   4. Biologics (e.g., interferon, interferon inducers, or immunomodulators); 28 days
   5. Glucocorticosteroids; 28 days
   6. Anti-metabolites (e.g., methotrexate); 28 days
   7. Vismodegib; 180 days
   8. Known photosensitizing medications or CYP3A inducers/inhibitors; 28 days
6. Any use of the following topical therapies within the specified period, or unwilling to meet the following washouts, prior to the Baseline visit and while on study, or in a proximity to any DPNTL, that in the Investigator's opinion could interfere with the investigational product study treatment applications or the study assessments:

   1. Laser, light or other energy-based therapy [e.g., intense pulsed light (IPL), photo-dynamic therapy (PDT)]; 180 days
   2. Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-flurouracil, or ingenol mebutate; 60 days
   3. Retinoids; 28 days
   4. Microdermabrasion or superficial chemical peels; 14 days
   5. Glucocorticosteroids or antibiotics; 14 days
7. Occurrence or presence of any of the following within the specified period prior to the Baseline visit on or in the proximity of any DPNTL that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   1. Cutaneous malignancy; 180 days
   2. Sunburn; currently
   3. A pre-malignancy (e.g., actinic keratosis); currently
   4. Body art (e.g., tattoos, piercing, etc.); currently
8. History of sensitivity to any of the ingredients in the investigational product.
9. Any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or other condition(s) (e.g., sunburn, excessive hair, open wounds, lupus, photosensitive disorders etc.) that, in the opinion of the Investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
10. Participation in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to the Screening visit.
11. History of hypertrophic scarring or keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of all DPNTLs that achieve clearance (DPNLA score of 0) | Through week 16
  The DPNLA is an Investigator assessment of DPN-variant of SK lesion severity based on presence of DPN and visibility of the DPN lesion.
  0 Clear: no visible DPN lesion
  1. Near Clear: a slightly visible DPN lesion; lesion may be macular
  2. Small: a visible DPN lesion with a diameter of less than 3 mm
  3. Large: a visible DPN lesion that is elevated with a diameter > 3mm
Assessment of the severity of the Application Site Reactions and review of adverse events | Through week 16
  Signs and Symptoms of Application Site Reactions (ASRs) include pain, burning, stinging, pruritus, erythema, edema, exudation, erosion/ulceration, hyperpigmentation, and hypopigmentation.

SECONDARY OUTCOMES:
Proportion of all DPNTLs achieving a DPNLA of 0 or 1 | Through week 16
  The DPNLA is an Investigator assessment of DPN-variant of SK lesion severity based on presence of DPN and visibility of the DPN lesion.
Time to DPNTLs achieving a DPNLA of 0 | Through week 16
  The DPNLA is an Investigator assessment of DPN-variant of SK lesion severity based on presence of DPN and visibility of the DPN lesion.
Percentage of subjects achieving clearance of all DPNTLs | Through week 16
Percentage of subjects achieving clearance of at least 60% of all DPNTLs | Through week 16
Percentage of all DPNTLs per subject achieving a DPNLA of 0 | Through week 16
  The DPNLA is an Investigator assessment of DPN-variant of SK lesion severity based on presence of DPN and visibility of the DPN lesion.
Percentage of all DPNTLs with a SSA (Subject's Self-Assessment) of 0 or 1 | Through week 16
  The SSA is a subject's self-reported assessment of DPN lesion severity based on presence and visible elevation of a DPN lesion. The SSA will be determined by all subjects for each DPNTL at all study visits from Visit 1/Screening to Visit 9/Last Visit
  0 No visible DPN lesion
  1. Mild: Slightly raised DPN lesion
  2. Moderate: Obviously raised DPN lesion
  3. Severe: Prominent DPN lesion
Percentage of all DPNTLs with a SSA of 0 | Through week 16
  The SSA is a subject's self-reported assessment of DPN lesion severity based on presence and visible elevation of a DPN lesion. The SSA will be determined by all subjects for each DPNTL at all study visits from Visit 1/Screening to Visit 9/Last Visit
  0 No visible DPN lesion
  1. Mild: Slightly raised DPN lesion
  2. Moderate: Obviously raised DPN lesion
  3. Severe: Prominent DPN lesion
Percent recurrence of all DPNTLs | Through week 16
Comparison of DPNTLs achieving DPNLA 0 at week 16 to baseline greatest diameter | Through week 16
Comparison of the percentage of DPNTLs/subject achieving DPNLA 0 at week 16 to number of enrolled DPNTLs/subject | Through week 16
Comparison of % clearance of DPNTLs at week 16 to onset, frequency, and severity of Application Site Reactions (ASRs) | Through week 16
Comparison of % clearance of DPNTLs at week 16 to subject satisfaction assessment score | Through week 16
Assess superiority of active over vehicle as measured by the subject satisfaction assessment score for their DPNTLs at week 16 | Through week 16
Dermoscopic diagnostic accuracy of DPNTLs, as confirmed by histology at week 16 | Through week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California, United States